CLINICAL TRIAL: NCT07009119
Title: Feasibility, Safety and Short-term Oncosurgical Outcome of Laparoscopic Pancreaticoduodenectomy for Malignancy: A Single Centre Experience
Brief Title: Laparoscopic Pancreaticoduodenectomy
Acronym: LPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1496/04/2025
Record Dates: First submitted 2025-05-20; First posted 2025-06-06 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer; Pancreatic Fistula; Periampullary Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Laparoscopic pancreaticoduodenectomy (Other): Laparoscopic pancreaticoduodenectomy:
  1. dissection
  2. reconstruction
  Interventions: Procedure: laparoscopic Pancreaticoduodenectomy

INTERVENTIONS:
Procedure: laparoscopic Pancreaticoduodenectomy — The patient is positioned in French position (right arm in, left arm abducted 90°), with a suprapubic area reserved for Pfannenstiel incision. A 6-port technique is used: sub-umbilical (12 mm), four semi-circular trocars (two 12 mm, two 5 mm), and a sub-xiphoid trocar for liver retraction. Laparoscopic pancreaticoduodenectomy (LPD) proceeds if no vascular invasion/metastasis is found. Key steps include Kocher's maneuver, vessel ligation (gastroepiploic, gastric, gastroduodenal), lymphadenectomy (stations 5-17), pancreatic neck transection, and jejunal division. Reconstruction involves duct-to-mucosa pancreaticojejunostomy (or invaginating if duct unfound), hepaticojejunostomy, and stapled gastrojejunostomy. Margins are examined post-resection. Harmonic scalpel/Ligasure and staplers are used.
  Other Names: LPD

SUMMARY:
Laparoscopic pancreaticoduodenectomy was first performed by Garner and Pomp in 1994. This is a technically difficult, time consuming and high rate of complication procedure. The reason is that duodenum and head of pancreas locate deeply in retroperitoneum and are surrounded by important structures such as inferior vena cava, abdominal aorta, superior mesenteric artery, superior mesenteric vein (SMV), portal vein (PV) and hepatic arteries. Injuring these structures during the surgery can lead to life-threatening complications. Moreover, doing anastomoses through laparoscopy, especially pancreatic anastomosis, is more difficult and takes more time than through open approach. The outcome of PD has improved over the last two decades due to advances in surgical techniques, anesthesia and perioperative care. Although studies from high volume centers demonstrate reduce in the operative mortality to less than 3%, the postoperative morbidity rate is still ranging from 30% to 60%. Laparoscopic surgery is being used increasingly as a less invasive alternative to traditional interventions for pancreatic resection. Laparoscopic pancreaticoduodenectomy (LPD) is a difficult procedure that has become increasingly popular. Nevertheless, comparative data on outcomes remain limited. In this prospective study, investigators evaluate the safety and feasibility of surgical and oncological outcomes of minimally invasive PD.

DETAILED DESCRIPTION:
Open pancreaticoduodenectomy (PD) was the standard treatment for a wide array of periampullary and pancreatic diseases including malignant and benign conditions. The outcome of PD has improved over the last two decades due to advances in surgical techniques, anesthesia and perioperative care . Although studies from high volume centers demonstrate reduce in the operative mortality to less than 3%, the postoperative morbidity rate is still ranging from 30% to 60%. Laparoscopic surgery is being used increasingly as a less invasive alternative to traditional interventions for pancreatic resection. Laparoscopic pancreaticoduodenectomy (LPD) is a difficult procedure that has become increasingly popular. Nevertheless, comparative data on outcomes remain limited despite several improvements in surgical devices and techniques that have allowed surgeons to approach the pancreas laparoscopically, laparoscopic PD remains challenging. LPD represents one of the most advanced abdominal operations owing to the necessity of a complex dissection and reconstruction. Recent reports note that complete laparoscopic PD including laparoscopic resection and reconstruction is both technically feasible and safe. In this prospective study, investigators evaluate the safety and feasibility of surgical and oncological outcomes of minimally invasive PD.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the curative treatment intent in accordance with clinical guidelines:

  * No evidence of metastasis.
  * Radiological non-involvement of superior mesenteric vein & portal vein.
  * Preserved fat planes between celiac axis, hepatic artery & superior mesenteric artery.
* Patients presenting with resectable pancreatic head cancer, cholangiocarcinoma, duodenal cancer and ampullary tumours who are fit for laparoscopic pancreaticoduodenectomy.

Exclusion Criteria:

* Unfit patients for surgery due to severe medical illness.
* Inoperable patients with distant metastases, including peritoneal, liver, distant lymph node metastases, and involvement of other organs.
* Irresectable tumors in diagnostic laparoscopy.
* Patients requiring left, central or total pancreatectomy or other palliative surgery.
* History of other malignant disease.
* Pregnant or breast-feeding women.
* Patients with serious mental disorders.
* Patients with vascular invasion and requiring vascular resection as evaluated by the multidisciplinary team team according to abdominal imaging data.
* Pancreatoduodenectomy for other diagnosis like cystic lesions, benign tumors or chronic calcific pancreatitis
* Patients with cirrhotic liver.
* Patients refused to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Assessment of Surgical Specimens | Assessed at the time of surgical specimen pathological evaluation (typically within 1-2 weeks post-surgery).
  Evaluation of the surgical specimens will include:
  * Number of lymph nodes harvested: Total count of lymph nodes excised and examined during surgery.
  * Resected margin status: Assessment of the presence or absence of tumor cells at the resection margins, classified as negative (R0), microscopic positive (R1), or macroscopic positive (R2).
  * Ratio of positive lymph nodes to total lymph nodes harvested: Proportion (%) calculated by dividing the number of histopathologically confirmed metastatic lymph nodes by the total number of lymph nodes retrieved.

SECONDARY OUTCOMES:
The rate of pancreatic fistula after pancreaticoduodenectomy | 4 weeks postoperative
  On or after the third postoperative day, the drain outflow of any detectable volume was treated as a pancreatic fistula with an amylase content larger than three times the upper normal serum amylase value
Operative time in minutes | From time of skin incision till time of skin closure
  Time spent in surgery
Intra-operative blood loss | day 0 (at the end of surgery)
  the amount of intra-operative blood loss (ml) at the end of surgery (d0): recorded by the anesthetist using a vacuum system.
Postoperative length of stay | up to 90 days
  the time from being admitted to hospital to discharge
Amount of intraoperative blood transfusion | From start of surgery of every participant till skin closure
  Amount of intraoperative packed red blood cell units transfused intraoperative
Length of postoperative surgical intensive care unit stay | From the date of admission to surgical intensive care unit after surgery to the date of discharge to ward or death whichever comes first, assessed up to 3 months .
  Length of postoperative surgical intensive care unit stay In days

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital , Minia University, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No